CLINICAL TRIAL: NCT00155012
Title: Clinical Application of 16-Detector Row Computed Tomography in Coronary Artery Disease
Brief Title: Clinical Application of MDCT in Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9361700491; NSC-93-2314-B-002-190
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-04

CONDITIONS: Coronary Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
1) Establish normal value for coronary calcium scoring in Taiwan. 2) Find out the relationship of coronary calcium deposition and coronary artery stenosis. Propose a clinical management guideline based on coronary calcium score. 3) Evaluate sensitivity/specificity of coronary CT angiography and the influence of coronary calcium score on coronary CT angiography. 4) Evaluate the clinical application of myocardial enhancement measurement.

DETAILED DESCRIPTION:
Computed tomography is evolving as a tool for noninvasive diagnosis of coronary artery disease. Coronary calcium deposition amount is an established independent coronary artery disease risk factor. However, coronary artery stenosis seldom occurred in the same location as calcium deposition. With the advent of 16-detector-row multislice spiral CT, direct visualization of coronary artery is possible. But it remains a great challenge to obtain diagnostic quality image in the beating heart. Small distal vessels may not be adequately visualized. Artifacts from severe calcification or coronary stent may render diagnosis difficult. The clinical implication of coronary calcium score, indication of coronary CT angiography and myocardial enhancement measurement should be further studied. The purposes of this study are: 1) Establish normal value for coronary calcium scoring in Taiwan. 2) Find out the relationship of coronary calcium deposition and coronary artery stenosis. Propose a clinical management guideline based on coronary calcium score. 3) Evaluate sensitivity/specificity of coronary CT angiography and the influence of coronary calcium score on coronary CT angiography. 4) Evaluate the clinical application of myocardial enhancement measurement.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease admitted for coronary angiography

Exclusion Criteria:

* Heart failure, irregular heart rate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-08; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Wen-jeng Lee, M.D., Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan